CLINICAL TRIAL: NCT04563377
Title: A Phase 1/2a Open Label Trial to Assess Safety and Immunogenicity of Candidate T-cell Vaccines ChAdOx1.HTI and MVA.HTI Given Sequentially to Healthy HIV-1/2 Negative Adult Volunteers in Oxford, UK
Brief Title: Safety and Immunogenicity of Candidate HIV Vaccines Given Sequentially
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HIV-CORE 0051
Record Dates: First submitted 2020-09-10; First posted 2020-09-24 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ChAdOx1.HTI and MVA.HTI vaccination (Experimental): 1x dose of ChAdOx1.HTI at 5 x 10^10 vp
  1x dose of MVA.HTI at 2 x 10^8 pfu
  Interventions: Biological: ChAdOx1.HTI and MVA.HTI

INTERVENTIONS:
Biological: ChAdOx1.HTI and MVA.HTI — ChAdOx1. HTI dose 5 x 10^10 vp MVA.HTI dose 2 x 10^8 pfu

SUMMARY:
The primary object of the study is to assess the safety profile of candidate vaccines ChAdOx1.HTI and MVA.HTI administered sequentially in healthy HIV-1/2 negative adult volunteers.

In addition, the study will assess the immune responses generated of the candidate vaccines ChAdOx1.HTI and MVA.HTI administered sequentially in healthy HIV-1/2 negative adult volunteers.

10 healthy, HIV-negative adult volunteers will receive one vaccination of CHAdOx1.HTI followed by a one vaccination of MVA.HTI 8 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-65 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their GP
* Women of child-bearing potential (defined as a fertile woman post-menarche until post-menopausal, unless permanently sterile due to total abdominal hysterectomy, bilateral salpingectomy and bilateral oophorectomy) agree to practice continuous effective contraception during the study and test negative for pregnancy on the day(s) of screening and vaccination
* For sexually active men, willingness to use barrier methods for the purposes of contraception from screening until 4 months after the last vaccination
* Agreement to refrain from blood donation during the course of the study
* In the opinion of the Investigators, the volunteer has understood the information provided. Written informed consent must be given before any study-related procedures are performed
* Willing to undergo HCV, HBV, syphilis and HIV testing, counselling and receive test results

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Receipt of a recombinant simian adenoviral vaccine prior to enrolment
* Planned receipt of another adenoviral vectored vaccine within 90 days after the vaccination with the ChAdOx1.HTI IMP
* Receipt of any investigational HIV-1/2 vaccine within the last 6 years
* Receipt of live attenuated vaccine within the previous 60 days or planned receipt within 60 days after vaccination with the IMP
* Receipt of other vaccine, including influenza vaccine, within the previous 14 days or planned receipt within 14 days after vaccination with the IMP
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV-1/2 infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis in relation to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin)
* History of serious psychiatric condition likely to affect participation in the study
* Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Reported high-risk behaviour for HIV-1/2 infection. High-risk behaviour for HIV-1/2 infection is defined as follows. Within the previous 12 months the volunteer has:

  * Had unprotected vaginal or anal sex with a known HIV-1/2-infected person or a casual partner (i.e., no continuing, established relationship)
  * Engaged in sex work for money or drugs
  * Used injection drugs
  * Acquired one of the following sexually transmitted infection: chlamydia, gonorrhoea and syphilis.
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Untreated Syphilis: Treponemal IgG/IgM and positive RPR/TPPA AND no documentation of adequate treatment
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Collection of data on adverse events. | Up to 8 months
  Occurrence of reactogenicity signs and symptoms for 7 days following vaccination Change from baseline for safety laboratory measures Occurrence of serious adverse events during the whole study duration

SECONDARY OUTCOMES:
Assessing the immunogenicity of the ChAdOx1.HTI and MVA.HTI vaccines administered sequentially | Up to 8 months
  Proportion of participants that develop T cell responses to HTI-encoded regions as determined by IFN-γ ELISPOT assay

CONTACTS AND LOCATIONS:
Overall Officials: Paola Cicconi, Principal Investigator — Dr Paola Cicconi
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No